CLINICAL TRIAL: NCT01298804
Title: Preventing Maternal Depression In Head Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Head Start and Early Head Start Programs in Action for Boston Community Development Incorporated (Unknown)
Responsible Party: Principal Investigator, Michael Silverstein, Associate Professor of Pediatrics, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH091871 (NIH)
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Problem Solving Education (Experimental)
  Interventions: Behavioral: Problem Solving Education and Activated Referral to Care
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Problem Solving Education and Activated Referral to Care — The intervention represents an integrated identification and intervention system based on the evidence-based construct of screening, brief intervention, and referral to treatment (SBIRT). Within the comprehensive case management services of Head Start, eligible women will be randomized to receive either usual care or the Head Start-based intervention. In our intervention, mothers at risk for depression will receive a problem-solving intervention; depression symptom monitoring; and an "Activated" referral to more definitive services for those who have worsening symptoms over time.
  Arms: Problem Solving Education

SUMMARY:
Maternal depression disproportionately affects low-income and minority women, and has profound negative impacts on their children. The investigators are conducting a randomized trial of a systems approach to identify mothers at risk for depression in Head Start - a federally funded early learning program for children of low-income families - and to provide an on-site intervention to prevent or alleviate depressive symptoms; improve functioning; and, where appropriate, proactively link mothers to more definitive mental health services.

DETAILED DESCRIPTION:
This study is one component of a series of studies that aims to develop a comprehensive system of maternal depression prevention and management within Head Start. In our March 2014 review of the CT.gov protocol, we synchronized it with our institution's IRB protocol, which had been modified based on how the individual studies within this series relate to one another. Specifically, the original IRB protocol combined two studies into one: a 'main' depression prevention trial (n=230, R01MH091871), and a small adjunct pilot aimed at referring those with symptoms of major depression to further care (n=60). Thus, the original CT.gov protocol included subjects both at risk for depression and with symptoms consistent with major depression. When the latter pilot study subsequently received external funding, we separated the two studies into two IRB protocols, and thus have adjusted our CT.gov protocol to the appropriate sample size of 230, and indicated symptoms of major depression as an exclusion criterion for the prevention trial. Because Major Depressive Episode was inadvertently listed as a primary outcome measure for the prevention trial (and PTSD and Anxiety as secondary outcome measures), we have removed them as such and listed it under 'other' outcomes, thereby aligning the CT.gov protocol with the statistical analysis plan of the original grant application and IRB protocol. Lastly, we corrected administrative errors in the study's projected end date and masking design.

ELIGIBILITY:
Inclusion Criteria:

* Family enrolled in Head Start, and child expected to attend Head Start activities for at least 6 months of the 12-month follow-up period.
* Family without imminent plans to relocate
* Mother is comfortable in English or Spanish.
* Parent/guardian who has a child that attends Head Start
* Child attending Head Start and is between the ages 0-5
* Screen positive to 2-question depression screener (PHQ2), or have a past history of depression
* Ability to provide informed consent.
* Not suicidal

Exclusion Criteria:

* High suicidal ideation
* Cognitive limitation
* Psychosis
* No known risks for depression
* Symptoms reflecting major depressive episode

Ages: 15 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 230 (Actual)
Dates: Start 2011-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Depression Symptoms | 2 months
  QIDS
Depression Symptoms | 4 months
  QIDS
Depression Symptoms | 6 months
  QIDS
Depression Symptoms | 8 months
  QIDS
Depression Symptoms | 10 months
  QIDS
Depression Symptoms | 12 months
  QIDS
Problem Solving Skills | 6 months
  Social Problem Solving Inventory
Problem Solving Skills | 12 months
  Social Problem Solving Inventory

SECONDARY OUTCOMES:
Social functioning | 6 months
  Social Adjustment Scale- Self-report
Parent functioning/stress | 6 months
  Parenting Stress Index; Perceived Stress Index
Head Start attendance | 12 months
  Head Start records, analyzed as monthly absence rates
Receipt of Mental Health Services | 12 months
Social functioning | 12 months
  Social Adjustment Scale- Self-report
Parent functioning/stress | 12 months
  Parenting Stress Index, Perceived Stress Index
Child Behavior | 6 months
  Teacher Version of Social Skills Rating System

OTHER OUTCOMES:
Major Depressive Episode | 12 months
  SCID Interview
Post Traumatic Stress Disorder | 12 months
  SCID Interview
Anxiety | 12 months
  SCID Interview

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverstein, MD, MPH, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - ABCD Head Start, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Silverstein M, Cabral H, Hegel M, Diaz-Linhart Y, Beardslee W, Kistin CJ, Feinberg E. Problem-Solving Education to Prevent Depression Among Low-Income Mothers: A Path Mediation Analysis in a Randomized Clinical Trial. JAMA Netw Open. 2018 Jun 1;1(2):e180334. doi: 10.1001/jamanetworkopen.2018.0334. PMID 30646083
- [Derived] Silverstein M, Diaz-Linhart Y, Cabral H, Beardslee W, Broder-Fingert S, Kistin CJ, Patts G, Feinberg E. Engaging Mothers With Depressive Symptoms in Care: Results of a Randomized Controlled Trial in Head Start. Psychiatr Serv. 2018 Nov 1;69(11):1175-1180. doi: 10.1176/appi.ps.201800173. Epub 2018 Sep 26. PMID 30256184
- [Derived] Silverstein M, Diaz-Linhart Y, Cabral H, Beardslee W, Hegel M, Haile W, Sander J, Patts G, Feinberg E. Efficacy of a Maternal Depression Prevention Strategy in Head Start: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Aug 1;74(8):781-789. doi: 10.1001/jamapsychiatry.2017.1001. PMID 28614554